CLINICAL TRIAL: NCT04243213
Title: "Pilot Study: Effects of Vibration on Postoperative Early Mobilization of Cardiac Surgery Patients"
Acronym: CardioVIB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Graz (Other)
Responsible Party: Principal Investigator, Nandu Goswami, Assoz. Prof. Dr., Medical University of Graz
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CardioVIB
Record Dates: First submitted 2020-01-20; First posted 2020-01-28 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Cardiovascular Risk Factor; Frailty
Keywords: early mobilisation after hospitalisation
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Intervention Model Description: Through a random selection process, the patients are divided into three groups of 10 patients each and receive the following treatment in addition to standard clinical physiotherapy:
  A: Intervention group I receives a unit of 10 minutes daily on the vibrating plate with an upright posture of 15 ° postoperatively from the 2nd to the 7th day B: Intervention group II is positioned postoperatively from day 2 to day 7 for 15 minutes at 15 degrees, but without vibration C: The control group only receives standard physiotherapy and no further treatments
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Vibration Group (Experimental): Intervention group I receives a unit of 10 minutes daily on the vibrating plate with an upright posture of 15 ° postoperatively from the 2nd to the 7th day
  Interventions: Other: Vibration Plate; Other: Tilt at 15°; Other: Standard hospital mobilization
- 15° Tilt Group (Experimental): Intervention group II is positioned postoperatively from day 2 to day 7 for 15 minutes at 15 degrees, but without vibration
  Interventions: Other: Tilt at 15°; Other: Standard hospital mobilization
- Control Group (Placebo Comparator): The control group only receives standard physiotherapy and no further treatments
  Interventions: Other: Standard hospital mobilization

INTERVENTIONS:
Other: Vibration Plate — Vibration at 15° tilt, which means the patients partly use their own body weight (resistive vibration exercise).
  Arms: Vibration Group
Other: Tilt at 15° — To compare if a possible effect derives from the vibration or the tilting only, a second group was added who will only receive 10 min of 15° tilt without the vibration.
  Arms: 15° Tilt Group; Vibration Group
Other: Standard hospital mobilization — early mobilization of patients 24h post surgery, done routinely, and physiotherapy this is done routinely in all patients

SUMMARY:
The rapid mobilization of cardiac surgery patients within the first 48 postoperative hours in the intensive care unit is common practice and decisive for the outcome, especially in this group (over 65 years). If sitting on the edge of the bed was successful, a standing attempt is usually made. Both can be accompanied by blood pressure dysregulations in the sense of hypotensive phases as well as dizziness. Postural control is the ability of the body to balance an upright body position under the influence of gravity.The aim of the study is to investigate whether training with the Galileo device by means of vibration on the soles of the feet and / or by changing the position to 15 ° can improve the postural control and thus the postoperative mobilization of patients.

DETAILED DESCRIPTION:
The aim of this study is to determine whether vibrations on the sole of the foot accelerate mobilization after cardiac surgery. Preliminary studies show that the mechanisms of cardiovascular regulation in the event of changes in position, e.g. when getting up from the lying position, can be positively influenced by vibration treatments on the soles of the feet, if at the same time a small part of the body weight is shifted to the soles of the feet. In the early phase after the operation, you may feel dizzy when you get up, which creates uncertainty in the patient, which in turn delays further mobilization.The sole of the foot vibrations and various measurements of the cardiovascular regulation are carried out in this study.

This study is carried out by the clinical department for cardiac surgery together with the chair of physiology at the Medical University of Graz. Thirty patients will participate in this study. Through a random selection process, the patients are divided into three groups of 10 patients each and receive the following treatment in addition to standard clinical physiotherapy:

A: Intervention group I receives a unit of 10 minutes daily on the vibrating plate with an upright posture of 15 ° postoperatively from the 2nd to the 7th day B: Intervention group II is positioned postoperatively from day 2 to day 7 for 10 minutes at 15 degrees, but without vibration C: The control group only receives standard physiotherapy and no further treatments

Standard physiotherapy consists of the patient trying to stand up together with the physiotherapist from the intensive care bed or IMC bed. The participation in this clinical trial will take approximately 60 minutes per appointment. This consists of 20-25 minutes for attaching the electrodes, 15 minutes for the "sit-to-stand test" and 15-20 minutes for the survey (filling out the questionnaires). At the beginning of the study or before the operation (OP), questionnaires are used to determine whether you have an increased risk of falling and whether you are frail. These questionnaires will be carried out by trained employees together with you during the initial measurement, upon discharge and after about 3 months.

To measure the cardiovascular regulation during changes in position, a sit-up test is carried out. Values such as blood pressure and cardiac output (Task Force Monitor), muscle activity on the calf over the skin and vascular reaction in the calf over the skin, and blood flow to the brain are measured with a Ultrasound device included. All methods used are non-invasive (that is, only adhesive electrodes are used on the skin and no needles or syringes, there is no blood draw in this measurement) and not painful. The patient will be asked to participate in such a sit-up test (from supine/lying position to standing upright) at a total of 5 measuring dates. In total the patient will be given two blood pressure cuffs, one on the right upper arm, the second on the left middle finger. To measure the ECG and other cardiovascular values, 8 electrodes are attached to your upper body. In addition there are 3 adhesive electrodes on the calves for measuring the muscles. No additional blood tests are carried out as part of the tests. The results of your routine blood tests will be included in the study.

All measurements from the patients in group A-C are compared to determine whether training with the vibration exercise leads to faster mobilization after cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients who undergo heart surgery: aortic valve replacement or elective coronary bypass

Exclusion Criteria:

* Euroscore II > 8
* patients with a postop. delirium on day 2 (drug treatment)
* Patients who require higher-dose catecholamines 48h post surgery (norepinephrine over 0.05-0.1 micrograms / kg body weight, suprarenin over 0.05-0.1 micrograms / kg body weight, Dobutrex over 5 micrograms / kg body weight)
* existing thrombosis

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Cardiopostural Control (heart rate) | changes comparing at following time-points: pre surgery + post surgery (24 hours, 7 days and 3 months)
  Changes in heart rate during sit-to-stand test before and after surgery as well as after rehabilitation (3 months follow up)
Cardiopostural Control (systolic blood pressure) | changes comparing at following time-points: pre surgery + post surgery (24 hours, 7 days and 3 months)
  Changes in systolic blood pressure during sit-to-stand test before and after surgery as well as after rehabilitation (3 months follow up)
Cardiopostural Control (diastolic blood pressure) | changes comparing at following time-points: pre surgery + post surgery (24 hours, 7 days and 3 months)
  Changes in diastolic blood pressure during sit-to-stand test before and after surgery as well as after rehabilitation (3 months follow up)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Graz, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: Undecided